CLINICAL TRIAL: NCT02095574
Title: Disposition of [14C] ABT-199 in Subjects With Relapsed or Refractory Non-Hodgkin's Lymphoma (NHL) Following a Single Oral Dose Administration
Brief Title: A Pharmacokinetic Study to Access How the Body Absorbs and Removes ABT-199 in Adults With Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: This study will now be conducted in healthy volunteers.
Sponsor: AbbVie (Industry)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: M13-363
Record Dates: First submitted 2014-01-28; First posted 2014-03-26 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Relapsed/Refractory Non-Hodgkin's Lymphoma
Keywords: GDC-0199; ADME; Relapsed; Refractory; ABT-199; Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Recurrence | interventions — venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]ABT-199 (Experimental): Subjects with relapsed or refractory Non-Hodgkin's Lymphoma
  Interventions: Drug: [14C]ABT-199 (GDC-0199)

INTERVENTIONS:
Drug: [14C]ABT-199 (GDC-0199) — [14C]ABT-199 will be administered as a single oral administration

SUMMARY:
A pharmacokinetic study to access how the body absorbs and removes ABT-199 in adults with Non-Hodgkin's Lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have relapsed or refractory disease.
2. Subject must have histologically documented diagnosis of non-hodgkin's lymphoma as defined by a B-cell neo-plasm in the World Health Organization (WHO) classification scheme except as noted in exclusion criteria.
3. Subject has an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.
4. Subject has adequate bone marrow (independent of growth factor support per local laboratory reference range).
5. Subject has adequate coagulation, renal and hepatic function.

Exclusion Criteria:

1. Subject has been diagnosed with Post-Transplant Lymphoproliferative Disease (PTLD), Burkitt's lymphoma, Burkitt-like lymphoma, lymphoblastic lymphoma/leukemia, chronic lymphocytic leukemia (CLL), mantle cell leukemia (MCL), or small lymphocytic lymphoma (SLL).
2. Subject has undergone an allogeneic stem cell transplant.
3. Subject is receiving combination anti-retroviral therapy for human immunodeficiency virus (HIV) (due to potential drug-drug interactions, as well as the potential for increased risk of opportunistic infections).
4. Subject has a significant history of renal, neurologic, psychiatric, endocrinologic, metabolic, immunologic, cardiovascular, or hepatic disease within 6 months that in the opinion of the Investigator would adversely affect his/her participation in this study.
5. Subject has active peptic ulcer disease or other hemorrhagic esophagitis/gastritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of ABT-199 and [14C]ABT-199 | For approximately 9 days following a single oral dose of [14C]ABT-199
Time to Cmax (Tmax) for ABT-199 and [14C]ABT-199 | For approximately 9 days following a single oral dose of [14C]ABT-199
Area Under the Time curve (AUC) for ABT-199 and [14C]ABT-199 | For approximately 9 days following a single oral dose of [14C]ABT-199
  The area under the exposure-time curve from time zero to Day 9 and time zero extrapolated to infinite time for single dose of [14C]ABT-199

SECONDARY OUTCOMES:
Number of subjects with adverse events | At each visit (daily for approximately the first 9 days)
  Adverse event monitoring, lab test assessment, physical exam and vital signs will be evaluated throughout the study.
Percentage of subjects with adverse events | At each visit (daily for approximately the first 9 days)
  Adverse event monitoring, lab test assessment, physical exam and vital signs will be evaluated throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Justin L Ricker, MD, Study Director — AbbVie